CLINICAL TRIAL: NCT06576219
Title: 'My Life is Music' Group Therapy Model - a Feasibility Study for Adolescents With Persistent Pain
Acronym: PedPainMusic
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Reetta Sipilä, PhD, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/564/2024
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Pain
Keywords: Pediatric Pain; Music Therapy; Group Therapy; Music Intervention; Persistent Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Behavioral: Group Music Therapy

INTERVENTIONS:
Behavioral: Group Music Therapy — My Life Is Music group therapy model

SUMMARY:
The aim of this multi-method feasibility study is to learn if a group therapy model using music can be applied in the treatment of adolescents with persistent pain. We are interested how the patients find participating in the group therapy as part of their rehabilitation and if the patient´s experience of music changes during the therapy process.

ELIGIBILITY:
Inclusion Criteria:

* persistent pain (3 months)
* fluency in finnish language

Exclusion Criteria:

- a psychiatric illness that significantly impairs functioning

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interviews | 12 weeks
  Patients and their parents
Patient Diaries | Weekly entries for 8 weeks during intervention
  patient's experiences on group therapy and music

SECONDARY OUTCOMES:
PROMIS Pediatric Profile | Baseline, 12 weeks
Music Questionnares | Baseline, 12 weeks
  B-MMR and BMRQ
Feedback Informed Treatment (FIT) | Baseline, weekly entries for 8 weeks during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- New Children´s Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided